CLINICAL TRIAL: NCT00861419
Title: An Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 386 With AMG 706, AMG 386 With Bevacizumab, AMG 386 With Sorafenib, and AMG 386 With Sunitinib in Adult Patients With Advanced Solid Tumors
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 386 When Used in Combination With AMG 706, Bevacizumab, Sorafenib, or Sunitinib.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050170
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Advanced Solid Tumors
Keywords: AMG 386; AMG 706; Bevacizumab; Sorafenib; Angiogenesis Inhibitors; Combination Therapy; Peptibody; Sunitinib
MeSH Terms: interventions — Sorafenib; motesanib diphosphate; trebananib; Sunitinib; Bevacizumab

ARMS (8):
- D (Experimental): 3 mg/kg AMG 386 IV (QW) / 125 mg AMG 706 PO (QD)
  Interventions: Drug: AMG 706; Drug: AMG 386
- A (Experimental): 3 mg/kg AMG 386 IV (QW) / 15 mg/kg bevacizumab IV (Q3W)
  Interventions: Drug: Bevacizumab; Drug: AMG 386
- B (Experimental): 3 mg/kg AMG 386 IV (QW) / 75 mg AMG 706 PO (QD)
  Interventions: Drug: AMG 706; Drug: AMG 386
- E (Experimental): 3 mg/kg AMG 386 IV (QW) / 400 mg sorafenib PO (BID)
  Interventions: Drug: Sorafenib; Drug: AMG 386
- H (Experimental): 10 mg/kg AMG 386 IV (QW) / 50 mg sunitinib PO (QD - 4 weeks on/2 weeks off)
  Interventions: Drug: AMG 386; Drug: Sunitinib
- G (Experimental): 3 mg/kg AMG 386 IV (QW) / 50 mg sunitinib PO (QD - 4 weeks on/2 weeks off)
  Interventions: Drug: Sunitinib; Drug: AMG 386
- C (Experimental): 10 mg/kg AMG 386 IV (QW) / 15 mg/kg bevacizumab IV (Q3W)
  Interventions: Drug: AMG 386; Drug: Bevacizumab
- F (Experimental): 10 mg/kg AMG 386 IV (QW) / 400 mg sorafenib PO (BID)
  Interventions: Drug: Sorafenib; Drug: AMG 386

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg PO (BID)
  Other Names: Nexavar
  Arms: E; F
Drug: AMG 706 — AMG 706 125 mg PO (QD)
  Other Names: Motesanib Diphosphate
  Arms: D
Drug: AMG 706 — AMG 706 75 mg PO (QD)
  Other Names: Motesanib Diphosphate
  Arms: B
Drug: AMG 386 — AMG 386 10 mg/kg IV (QW)
  Arms: C; F; H
Drug: Sunitinib — Sunitinib 50 mg PO (QD)
  Other Names: Sutent
  Arms: G; H
Drug: Bevacizumab — Bevacizumab 15mg/kg IV Q3W
  Other Names: Avastin
  Arms: A; C
Drug: AMG 386 — AMG 386 3 mg/kg IV (QW)
  Arms: A; B; D; E; G

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of AMG 386 when used in combination with AMG 706, bevacizumab, sorafenib, or sunitinib and that at least one dose level from each combination will be safe and well tolerated.

AMG 386 is a man-made medication that is designed to stop the development of blood vessels in cancer tissues. Cancer tissues rely on the development of new blood vessels, a process called angiogenesis, to obtain a supply of oxygen and nutrients to grow.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years old.
* Subjects must have a pathologically documented, and definitively diagnosed, advanced solid tumor that is refractory to standard treatment, for which no standard therapy is available, or for subjects who refuse standard therapy.
* Subjects enrolling in arms E & F and G & H must have pathologically documented and definitively diagnosed advanced renal cell carcinoma.
* Measurable disease or evaluable (non-measurable) disease per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status up to 2.
* Subjects must be able to self-administer AMG 706 (arms B and D) or sorafenib (arms E and F) on an empty stomach (fasting for 1 hour before and 1 hour postdose) once daily for AMG 706 or twice daily for sorafenib. Subjects enrolling in arms G and H must be able to self-administer sunitinib once daily.

Exclusion Criteria:

* History of lymphoma or leukemia.
* Symptomatic or untreated central nervous system metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and corticosteroids.
* Subjects with head and neck cancer.
* Subjects with lung squamous cell tumors or with large central (located adjacent to or within the hilum or mediastinum) tumor lesions ≥ 3 centimeters, regardless of histology
* For arms A and C: Subjects with ovarian cancer.
* History of arterial or venous thrombosis or pulmonary embolism within 1 year before enrollment; history of bleeding diathesis.
* Cardiovascular events within 1 year before enrollment, such as myocardial infarction, unstable/severe angina, coronary/peripheral artery bypass graft, unstable cardiac arrhythmia requiring medication, symptomatic congestive heart failure (New York Heart Association >class II), cerebrovascular accident or transient ischemic attack.
* For arms G and H: LVEF ≤ 45%, heart rate < 50 / min.
* Chronic uncontrolled hypertension [diastolic > 85 mmHg; systolic >145 mmHg].
* History of pulmonary hemorrhage or gross hemoptysis within 6 months before enrollment.
* History of significant GI surgery or disease, which would impair absorption.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Active infection within 2 weeks before enrollment.
* Subject known to have tested positive for HIV.
* Subject known to have chronic hepatitis (e.g., hepatitis B or hepatitis C).
* Coumarin anticoagulants including warfarin, at doses greater than 2 mg/day. The concurrent use of low molecular weight heparin or low dose warfarin (ie, ≤ 2 mg daily for prophylaxis against central venous catheter thrombosis is acceptable.
* Treatment with anti-cancer therapy within 30 days before study day 1 (treatment with bevacizumab within 42 days before study day 1) unless prior written approval is received from the sponsor
* Hormonal anti-tumor therapy within 30 days before enrollment. Does not include hormones for non-cancer related conditions (eg, insulin for diabetes, HRT) or the use of gonadotropin-releasing hormone (GnRH) agonists for prostate cancer
* Therapeutic or palliative radiation therapy within 2 weeks before enrollment
* Prior treatment with AMG 386
* Prior radiation therapy to the abdomen
* For arms A, B, C, and D: prior treatment with bevacizumab, sorafenib, sunitinib, or investigational agents known to directly inhibit the functions of vascular endothelial growth factor, vascular endothelial growth factor receptors, angiopoietins, or angiopoietin receptors, unless prior written approval is received from the sponsor
* For arms E and F: prior treatment with sorafenib, unless prior written approval is received from the sponsor
* For arms G and H: prior treatment with sunitinib, unless prior written approval is received from the sponsor
* For arms E & F and G & H: treatment with bevacizumab within 42 days before study day 1, unless prior written approval is received from the sponsor
* Major surgery within 30 days before enrollment or recovering from prior surgery
* Subject who is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2005-12

PRIMARY OUTCOMES:
Safety including adverse events, clinically significant changes in laboratory results, ECG, and vital signs, to be measured throughout the study. Pharmacokinetic Profile of AMG 386 - blood levels of AMG 386 to be measured throughout the study.

SECONDARY OUTCOMES:
Response based on biomarker, anti-AMG 386 antibody formation and tumor response measure by RECIST. | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Hong DS, Gordon MS, Samlowski WE, Kurzrock R, Tannir N, Friedland D, Mendelson DS, Vogelzang NJ, Rasmussen E, Wu BM, Bass MB, Zhong ZD, Friberg G, Appleman LJ. A phase I, open-label study of trebananib combined with sorafenib or sunitinib in patients with advanced renal cell carcinoma. Clin Genitourin Cancer. 2014 Jun;12(3):167-177.e2. doi: 10.1016/j.clgc.2013.11.007. Epub 2013 Nov 13. PMID 24365125
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com